CLINICAL TRIAL: NCT05034874
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety and Efficacy of IXT-m200 in Treatment-Seeking Individuals With Methamphetamine Use Disorder
Brief Title: Multiple-Dose Study to Evaluate the Safety and Efficacy of IXT-m200
Acronym: OUTLAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis concluded planned study numbers combined with participant dropout rates were insufficient to meet primary endpoint.
Sponsor: InterveXion Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M200C-2201; U01DA055481 (NIH)
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-05

CONDITIONS: Methamphetamine-dependence; Methamphetamine Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IXT-m200 (Experimental): Anti-methamphetamine monoclonal antibody, dose levels of 1.5 and 3 g
  Interventions: Drug: IXT-m200
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IXT-m200 — IXT-m200 binds METH with high selectivity and affinity. The product contains a murine METH-binding variable region and the constant domains of a human immunoglobulin G (IgG) 2κ. This antibody isotype was chosen because of the lower risk of immune response compared to an IgG1 or IgG3. IXT-m200 targets METH, does not rely on binding to any endogenous target for its action, and has been well-tolerated in previous clinical studies.
  Arms: IXT-m200
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
This Phase 2 study will evaluate the safety and efficacy of monthly intravenous doses of IXT-m200 in treatment-seeking individuals with methamphetamine (METH) use disorder. The hypothesis are that following an initial relapse, IXT-m200 will reduce the occurrence of stimulant-positive saliva samples compared to placebo and improve the signs and symptoms of METH Use Disorder (MUD).

ELIGIBILITY:
Eligible participants will:

1. Be at least 18 years of age at the time of study consent;
2. Meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for Substance Use Disorder associated with methamphetamine;
3. Be treatment-seeking methamphetamine users with at least 1 methamphetamine or amphetamine positive specimen during the screening period;
4. Be able and willing to read, comprehend, and give Authorization for Use/Disclosure of Health Information (HIPAA) and informed consent;
5. Be willing to comply with study instructions and dosing, agree to make all appointments, and complete the entire course of the study;
6. Agree to use protocol-specified method(s) of birth control throughout study participation;
7. Agree to adhere to Lifestyle Considerations throughout study duration;
8. Have access to a smartphone or other device capable of supporting the study app;
9. Successfully complete app-based training program as evidenced by completion of at least 75% of daily drug use surveys and assigned saliva drug screens (two of which must be valid) in ≤30 days from the screening visit during the screening period.

Eligible participants will NOT:

1. Have current dependence, defined by DSM-5 criteria, on any psychoactive substance (i.e., opioids or benzodiazepines), other than methamphetamine or nicotine (any severity). Mild severity dependence on alcohol or marijuana is allowed;
2. Be currently taking certain other drugs and medications, including: "designer drugs" (e.g., 3,4-methylenedioxyMETH (MDMA, Ecstasy, Adam, XTC) and its N-dimethyl metabolite methylenedioxyamphetamine (MDA), anti-orexigenic drugs (including over-the-counter medications for weight loss), or be chronic users of phenethylamine compounds (e.g., phenylpropanolamine, ephedrine, pseudoephedrine, amphetamine, phentermine, phenmetrazine, methylphenidate, diethylpropion, and propylhexedrine);
3. Have a known contraindication or sensitivity to IXT-m200 based on known allergies to other monoclonal antibodies, any inactive ingredient of IXT-m200, or any other products required for the study procedures;
4. Have a history of severe allergy (rash, hives, breathing difficulty, etc) to any medications;
5. Have a history of allergic or environmental bronchial asthma within the past 3 years;
6. Have a current diagnosis of anorexia nervosa or bulimia disorder;
7. Have a history of unstable cardiovascular disease that is not adequately controlled at the time of eligibility determination;
8. Be mandated by the court to obtain treatment for methamphetamine-dependence where such mandate required the results of methamphetamine testing to be reported to the court;
9. Have positive saliva drug screens for psychoactive substances other than amphetamines at the screening visit;
10. Be expected to fail to complete the study protocol due to probable incarceration or relocation from the clinic area, or any clinically significant mental or physical illness within a 1-year prior, that would impact compliance with trial requirements;
11. Have clinically significant laboratory values (outside of normal limits). The following specified ranges are allowable:

    1. Liver function tests (total, direct, and indirect bilirubin, aspartate transaminase, alanine aminotransferase, gamma-glutamyl transferase, lactate dehydrogenase, and alkaline phosphatase) <3 times the upper limit of normal, and
    2. Kidney function tests (creatinine and BUN) <2 times the upper limit of normal;
12. Be considered to be at imminent risk of suicide or have a past-year history of a serious suicide attempt (defined as an attempt that results in or requires medical treatment) based on response to queries within eligibility screening about suicidal ideation and attempts;
13. Have an uncontrolled systemic disease or a medical condition that may increase the risk associated with study participation or administration of study treatment or that may interfere with the interpretation of study results;
14. Be currently participating or has participated within the last 30 days prior to the start of this study in a drug, device, or other interventional research study;
15. Be pregnant or lactating;
16. In the Investigator's or Sponsor's (or designee) opinion, be inappropriate for the study, including those believed to be attempting to enter the study primarily for financial gain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — InterveXion Therapeutics
Locations (9):
- United States (9):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Woodlands International Research Group, Little Rock, Arkansas
  - Artemis Institute for Clinical Research, San Diego, California
  - Pillar Clinical Research, Lincolnwood, Illinois
  - Midwest Clinical Research Center, Dayton, Ohio
  - InSite Clinical Research, DeSoto, Texas
  - HD Research, Houston, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Alpine Research, Clinton, Utah

IPD SHARING:
Plan to Share IPD: Yes
Final datasets are expected to contain IXT-m200 concentrations and immunogenicity results, METH use frequencies, Treatment Effectiveness Assessment scores, and safety data over time. No individually identifiable private information will be distributed.
Time Frame: These datasets will be available for distribution following submission to the FDA of the Clinical Study Report and publication. They will be available for 2 years after the initial publication.
Access Criteria: These datasets and associated documentation will be made available on CD by the Sponsor to requestors under a data sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology and not distributing to third parties; and (3) a commitment to destroying or returning the data after analyses are completed. Requests should be sent to intervexion@gmail.com.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were required to qualify for the study by complying with app-based drug testing assignments. In addition, one of the drug tests performed during the screening period must have been positive for methamphetamine (METH) to qualify.
Groups:
- IXT-m200: Anti-methamphetamine monoclonal antibody, dose level of 1.5 g
  IXT-m200: IXT-m200 binds METH with high selectivity and affinity. The product contains a murine METH-binding variable region and the constant domains of a human immunoglobulin G (IgG) 2κ. This antibody isotype was chosen because of the lower risk of immune response compared to an IgG1 or IgG3. IXT-m200 targets METH, does not rely on binding to any endogenous target for its action, and has been well-tolerated in previous clinical studies.
Period: Overall Study
Arm/Group | IXT-m200 | Placebo
Started | 41 | 20
Completed | 15 | 4
Not Completed | 26 | 16
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 18 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Skipped final visits, checked into rehab | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IXT-m200 | Placebo | Total
Number analyzed (Participants) | 41 | 20 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.13) | 46.8 (7.63) | 43.0 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 36
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 35 | 18 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 38 | 18 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Days per month of METH use [Number; unit: participants] — Participants were asked at Screening how many days in the past month they used methamphetamine. Responses were categorized as <18 days per month or ≥18 days per month.
  participants
    <18 days per month | 2 | 1 | 3
    ≥18 days per month | 39 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percent of 20 Weeks Abstinent From Stimulants Following a 4-week Grace Period
Description: The difference in group means between the IXT-m200 and placebo groups for the percent of 20 weeks abstinent from stimulants following a 4-week grace period as measured by saliva screens in treatment-seeking individuals with Methamphetamine Use Disorder. All observations will be used, regardless of whether a participant discontinued treatment early. All missing values will be imputed assuming the participant is not abstinent.
Time Frame: 20 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: percentage of 20 weeks abstinent
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 41 | 20
percentage of 20 weeks abstinent | 5.9 (17.33) | 4.3 (8.73)

2. Secondary Outcome: Change From Screening in Participant-rated Quality of Life as Measured by the Treatment Effectiveness Assessment at Week 13, 25, and 33.
Description: Treatment Effectiveness Assessment (TEA) asks questions in four domains with results ranging from 4-40 with higher scores representing a better outcome.
Time Frame: Weeks 13, 25, and 33
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 41 | 20
score on a scale
  Week 13 | 6.2 (8.67) | 4.6 (8.16)
  Week 25 | 7.3 (9.07) | 17 (9.09)
  Week 33 | 11 (9.32) | 13.5 (10.25)

3. Secondary Outcome: Proportion of Responders in Early Remission at Week 25 as Measured by DSM-5 Criteria
Description: A responder is defined as a participant who meets the definition of early remission, i.e., at least 3 months and <12 months without meeting DSM-5 criteria other than craving.
Time Frame: 25 weeks
Population: Intent to treat
Measure: Number; unit: percentage of responders
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 41 | 20
percentage of responders | 2.4 | 0

4. Secondary Outcome: Difference Between Groups in Clinical Global Impression of Change (CGIC) at Week 13, 25, and 33
Description: The CGIC asks clinicians to complete one statement with the result ranging from 1-7 with lower scores representing a better outcome.
Time Frame: Weeks 13, 25, and 33
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 41 | 20
score on a scale
  Week 13 | 3 (1.11) | 3 (0.87)
  Week 25 | 3.1 (0.89) | 2.3 (0.96)
  Week 33 | 2.7 (1.28) | 2 (0.82)

5. Secondary Outcome: Difference Between Groups in Patient Global Impression of Change (PGIC) at Week 13, 25, and 33
Description: The PGIC asks patients to complete one statement with the result ranging from 1-7 with lower scores representing a better outcome.
Time Frame: Weeks 13, 25, and 33
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 41 | 20
score on a scale
  Week 13 | 2.8 (1.22) | 3 (0.87)
  Week 25 | 3 (1.55) | 2.5 (1.29)
  Week 33 | 2.3 (1.39) | 1.8 (0.96)

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | IXT-m200 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/41 | 2/20
Other Adverse Events (participants affected / at risk) | 21/41 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IXT-m200 (N=41) | Placebo (N=20)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IXT-m200 (N=41) | Placebo (N=20)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovainal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increase (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to missing data leading to small numbers of participants analyzed. Participants did not submit drug tests as required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor requires an opportunity to review any proposed disclosure at least 60 days prior to disclosure. Potential modifications may be suggested. PI will delete any information identified as confidential by sponsor or defer to permit filing of any patent applications. First publication will be a joint publication by Sponsor involving all trial sites. PI may publish if joint manuscript not submitted within 12 months of completion of clinical study report or termination of the trial at all sites.

DOCUMENTS (3):
  • Study Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT05034874/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT05034874/SAP_001.pdf
  • Informed Consent Form (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT05034874/ICF_002.pdf